CLINICAL TRIAL: NCT04290481
Title: Oxygen Saturation and Perfusion Index Screening ın Neonates at High Altitude
Brief Title: Oxygen Saturation and Perfusion Index ın Neonates at High Altitude
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Kadir Şerafettin Tekgündüz, Associate Prof, Ataturk University
Other Study IDs: B.30.2.ATA.0.01.00/32
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Critical Congenital Heart Disease; High Altitude
MeSH Terms: conditions — Altitude Sickness | interventions — Oxygen Saturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: oxygen saturation and perfusion index screening — Oxygen saturation and perfusion index values that are measured by pulse oximeter is used for screening critical congenital heart disease.

SUMMARY:
Congenital heart diseases are among the most common congenital anomalies and occur with an incidence of approximately 8ınd12 / 1,000 live births worldwide. This figure does not cover minor lesions such as bicuspid aortic valves and small atrial or ventricular septal defects. Most of these defects do not need treatment or treatment is needed after infancy. Other defects are severe and usually require early treatment in the neonatal period. Critical congenital heart disease is defined as structural heart defects that are associated with hypoxia in the neonatal period and have significant morbidity and mortality potential in early life. Critical congenital heart disease is estimated to be ~3 in 1000 live births. It is estimated that 50% of congenital heart diseases are detected by prenatal ultrasound. Even if a standard neonatal examination is performed, 13 to 55% of patients with critical congenital heart disease can be discharged from the hospital without being diagnosed.

Screening of infants with non-invasive oxygen saturation measurement has been proposed as an adjunct to early detection of critical congenital heart disease.

The American Academy of Pediatrics, the American Cardiology Foundation and the American Heart Association have targeted 7 specific lesions for the pulse oximetry screening protocol: truncus arteriosus, transposition of the great arteries, tricuspid atresia, tetralogy of Fallot, total pulmonary venous return anomaly, hypoplastic left heart syndrome and pulmonary atresia.

The reference values of peripheral perfusion (PPI) index has been established for normal newborns between 1 and 120 h of age.

Lower PPI values than 0.70 may indicate illness. Including cut-off values for PPI in pulse-oximetry screening for duct dependent congenital heart disease is a promising tool for improving the detection of critical congenital heart disease with duct-dependent systemic circulation.

We aimed to investigate screening critical congenital heart disease and also to establish normal values of oxygen saturation and perfusion index at high altitude.

ELIGIBILITY:
Inclusion Criteria:

* The newborns delivered in Ataturk University Hospital and ≥34 weeks of gestational age were eligible for the study.

Exclusion Criteria:

* Outborn and premature babies (<34 weeks) were not included. Babies with a prenatal diagnosis of congenital heart disease were excluded.

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns with ≥34 weeks of gestational age
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Establishing threshold values for critical congenital heart disease screening at high altitude | Postnatal 24-48 hours
  We aim to explore whether oxygen saturation and perfusion index threshold values are different compared sea level or not.

SECONDARY OUTCOMES:
Establishing normal oxygen saturation and perfusion index values at high altitude | Postnatal 24-48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Medical Faculty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No